CLINICAL TRIAL: NCT04166643
Title: The Worksite Heart Health Improvement Project (WHHIP) + Function Focused Care (FFC)
Brief Title: Worksite Wellness Within Long-term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: American Heart Association (Other); Building Healthy Behaviors Across the Life Span Research Center (Unknown)
Responsible Party: Principal Investigator, Kelly Doran, associate professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00086939; 19TPA34830011 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2019-11-05; First posted 2019-11-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-11

CONDITIONS: Worksite Health Promotion; Lifestyle Risk Reduction; Cardiovascular Diseases; Occupational Stress; Healthcare Workers
MeSH Terms: conditions — Risk Reduction Behavior; Cardiovascular Diseases; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education only (Active Comparator): Education
  Interventions: Behavioral: Education only control
- WHHIP-PLUS and Function Focused Care (Experimental): Component I: Stakeholder Group Involvement:
  Component II: Environment Assessment:
  Component III: Organizational Changes To Reduce Job Stress:
  Component IV- Worker Health Behavior Change including function focused care interventions
  Interventions: Behavioral: WHHIP PLUS

INTERVENTIONS:
Behavioral: WHHIP PLUS — Worksite health promotion and occupational health and safety (total worker health)
  Arms: WHHIP-PLUS and Function Focused Care
Behavioral: Education only control — Education at the start of the project
  Arms: Education only

SUMMARY:
The goal of this proposed study is to test the feasibility and preliminary efficacy of worksite wellness program designed to reduce worker stress (job and personal) and improve cardiovascular disease among long-term care workers. We also aim to test if increasing wellness behaviors in staff will translate to increased wellness behaviors in residents due to positive role modeling.

DETAILED DESCRIPTION:
This is a cluster randomized control trial (initially intended to recruit 246 staff and 180 residents) implemented in six long-term care worksites. Three sites will be randomized to the WHHIP-PLUS & FFC and three sites will be randomized to the education-only.

The intervention occurs over 12 months and measures will be collected at three timepoints. We will test treatment fidelity as well as if our intervention improves Life's Simple 7 scores and reduces stress levels among long-term care workers and increases physical activity among residents.

ELIGIBILITY:
Staff inclusion criteria:

18 years or older; Able to understand and speak English; Employed by the facility; Passed the evaluation to sign consent

Resident inclusion criteria:

55 years or older; Able to understand and speak English; Resident of the facility; Passed the evaluation to sign consent

No exclusion criteria for staff or residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease risk | baseline, 6-months, 12-months
  Composite life simple 7 scores and individual scores from life simple 7 components (blood pressure, weight, cholesterol, blood sugar, tobacco exposure, diet, physical activity) for staff

SECONDARY OUTCOMES:
Short version of the Depression Anxiety Stress Scale-Stress- (DASS-S) | baseline, 6-months, 12-months
  Personal mood assessment tool, it can be scored as a composite mood score or three individual subscales, higher indicates more stress, 0-21 for each subscale or 0-63 for the composite for staff
Job strain model tool | baseline, 6-months, 12-months
  Tool to measure work environment for staff including job control (including decision authority [9 items, range 9-36] and skill discretion [6 items, range 6-24]), job demands (4 items, range 4-16), social support (6 items, range 6-24 ), and organizational justice (5 items, range 5-20). Lower scores are desired.

OTHER OUTCOMES:
Modified Nursing Assistant Self-efficacy for Restorative Care (NASERC) | baseline, 6-months, 12-months
  Tool to assess staff encouraging their patients to engage in heart healthy behaviors, range 0-36, higher means more self-efficacy for staff
Modified Nursing Assistant Outcome Expectations for Restorative Care (NAOERC) | baseline, 6-months, 12-months
  Tool to assess staff encouraging their patients to engage in heart healthy behaviors, range 0-44, higher means more outcome expectations for staff
Sleep | baseline, 6-months, 12-months
  Accelerometer for staff
Bioelectrical Impedance Analysis (BIA) | baseline, 6-months, 12-months
  Percent of body fat and muscle mass for staff
Modified Pittsburgh Sleep Quality Index | baseline, 6-months, 12-months
  Individual items on sleep hours and quality for staff
Barthel index | baseline, 6-months, 12-months
  Assesses functional independence for residents
Function focused care | baseline, 6-months, 12-months
  This tool is on observational check list that assesses long-term care staff and resident interactions for encouragement in function focused care (i.e., how staff engage or encourage residents to engage in physical activity). Staff are observed for about 30 minutes and scored (performed, not performed, not observed) on encouragement of function focused care for 19 typical care items such as bed mobility, ambulation in hallway.
3 word recall from mini-cog | baseline, 6-months, 12-months
  Stating 3 words to residents and asking them to recall them words.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Doran, PhD, RN, Principal Investigator — UMB
Locations (1):
- University of Maryland School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data
Time Frame: Once the study and preliminary analysis is complete (anticipated date 2025). Once published it will remain available
Access Criteria: open